CLINICAL TRIAL: NCT03791320
Title: Multicenter Validation of 3D-QCA Based FFR vs. Pressure Wire Based FFR: The FAST-II Study
Brief Title: Fast Assessment of STenosis Severity- FASTII Study
Acronym: FASTII
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Tokyo Medical University (Other); Centro Cardiologico Monzino (Other); Columbia University (Other); University Hospital Carl Gustav Carus (Other); University Hospital, Lille (Other)
Responsible Party: Principal Investigator, Joost Daemen, Principal Investigator, Erasmus Medical Center
Other Study IDs: FASTII Study: June 26, 2018
Record Dates: First submitted 2018-12-20; First posted 2019-01-02 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Coronary Artery Disease
Keywords: Fractional Flow Reserve; Coronary Physiology; 3D-QCA; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Vessel Fractional Flow Reserve — FFR measurement based on coronary angiography
  Other Names: 3D-QCA based FFR

SUMMARY:
The Multicenter FAST (Fast Assessment of STenosis severity) study is a prospective observational multicenter study designed to evaluate the diagnostic accuracy of offline 3D-QCA based FFR, using CAAS Workstation (Pie Medical Imaging, Maastricht, the Netherlands) in identifying hemodynamically significant coronary artery disease with pressure wire-based FFR (≤0.80) as the reference standard.

DETAILED DESCRIPTION:
The Multicenter FAST study is a prospective observational multicenter international study in which offline computation of vFFR is compared to conventional invasive, wire based FFR measurements. Pressure wire based FFR will be performed in patients with at least one intermediate coronary lesion at the discretion of the operator (typically defined as a coronary artery lesion with a diameter stenosis of 30-70% by visual assessment). A total of 3 two-dimensional angiography images, will be recorded and exported to the CAAS workstation 8.0 (Pie Medical Imaging, Maastricht, the Netherlands): two orthogonal views to create a 3D reconstruction of the coronary arteries and one view to ascertain the position of the FFR pressure wire. vFFR will be calculated automatically, by using the invasively measured aortic root pressure. vFFR measurements will be performed online by the different centers. In addition, all angiographic imaging data will be sent to an independent core laboratory (Cardialysis, Rotterdam, The Netherlands) for offline analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years
* indication procedure: stable, unstable angina or non-ST elevation acute coronary syndrome
* Diagnostic coronary angiography or PCI with an indication to perform re-PCI FFR assessment of at least one coronary artery lesion.

Exclusion Criteria:

* ST-elevation myocardial infarction (STEMI)
* Cardiogenic shock
* Severe hemodynamic instability
* Adenosine intolerance
* Lesions containing thrombus, left main lesions, grafts, arteries with collaterals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients ≥ 18 years presenting with stable or unstable angina or non-ST elevation acute coronary syndrome.
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of vFFR to identify FFR (≤0.8 or >0.8) calculated by corelab | 1 year
  The diagnostic accuracy of offline vFFR assessed by a blinded independent core laboratory to identify hemodynamically-significant coronary stenosis with FFR (≤0.8 or >0.8) as the reference standard.

SECONDARY OUTCOMES:
Diagnostic accuracy of vFFR to identify FFR (≤0.8 or >0.8) calculated by site/operator | 1 year
  The diagnostic accuracy of operator or cathlab technician calculated online vFFR to identify hemodynamically-significant coronary stenosis with FFR (≤0.8 or >0.8) as the reference standard.
Interobserver variability | 1 year
  3D-QCA based FFR (vFFR) will be calculated twice: by the operator/technician of different centers AND by an independent corelab (Cardoalysis). Correlation and agreement between these two measurements will be assessed in order to investigate the Inter-observer variability.

CONTACTS AND LOCATIONS:
Overall Officials: Joost Daemen, MD;PhD., Principal Investigator — Erasmus Medical Center
Locations (6):
- Columbia University Medical Center, New York, New York, United States
- CHU, Lille, France
- Herzzentrum Dresden, Dresden, Germany
- Centro Cardiologico Monzino, Milan, Italy
- Tokyo Medical University, Tokyo, Japan
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Individual participant data are needed for the final analysis which will be done by Erasmus MC.

REFERENCES:
- [Derived] Masdjedi K, Tanaka N, Van Belle E, Porouchani S, Linke A, Woitek FJ, Bartorelli AL, Ali ZA, den Dekker WK, Wilschut J, Diletti R, Zijlstra F, Boersma E, Van Mieghem NM, Spitzer E, Daemen J. Vessel fractional flow reserve (vFFR) for the assessment of stenosis severity: the FAST II study. EuroIntervention. 2022 Apr 22;17(18):1498-1505. doi: 10.4244/EIJ-D-21-00471. PMID 34647890